CLINICAL TRIAL: NCT04506034
Title: Is Lidocaine Patch as Effective as Intravenous Lidocaine in Pain and Illus Reduction After Laparoscopic Gynecologic Surgery? A Randomized Clinical Trial
Brief Title: Lidocaine Patch Versus Intravenous Lidocaine in Pain Relief After Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: aswu/277/7/18
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lidocaine patches (Experimental): for every port entry site from the three in ports of laparoscope, patients received three lidocaine patches 5% (Lidoderm® , Endo Pharmaceuticals, Chadds Ford, PA). Each patch measured 10 cm × 14 cm and contains (700 mg), was divided into two equal parts, six parts applied two of it around one port entry site that marked before sterilization and just before induction of anesthesia. The patches not changed until removed after return of bowel function or on the maximum at fifth postoperative day.
  Interventions: Drug: lidocaine patches
- IV lidocaine (Active Comparator): received i.v. lidocaine infusion after induction of anesthesia, 2 mg/min if body weight >70 kg or 1 mg/min if body weight <70 kg.
  Interventions: Drug: IV lidocaine
- IV saline infusion (Placebo Comparator): received i.v. saline infusion.
  Interventions: Drug: IV saline infusion

INTERVENTIONS:
Drug: lidocaine patches — for every port entry site from the three in ports of laparoscope, patients received three lidocaine patches 5% (Lidoderm® , Endo Pharmaceuticals, Chadds Ford, PA). Each patch measured 10 cm × 14 cm and contains (700 mg), was divided into two equal parts, six parts applied two of it around one port entry site that marked before sterilization and just before induction of anesthesia. The patches not changed until removed after return of bowel function or on the maximum at fifth postoperative day.
  Other Names: lidocaine patch
  Arms: lidocaine patches
Drug: IV lidocaine — received i.v. lidocaine infusion after induction of anesthesia, 2 mg/min if body weight >70 kg or 1 mg/min if body weight <70 kg.
  Other Names: lidocaine infusion
  Arms: IV lidocaine
Drug: IV saline infusion — received i.v. saline infusion.
  Other Names: placebo
  Arms: IV saline infusion

SUMMARY:
To evaluate the efficacy of lidocaine patch applied around wound in laparoscopic gynecologic surgery in reduction of postoperative pain and illus compared to intravenous lidocaine infusion and placebo.

DETAILED DESCRIPTION:
Postoperative pain after gynecologic surgery is a challenging problem associated with increased morbidity and cost. The inflammatory response to surgery plays a crucial rule in inducing postoperative illus. Systemic local anesthetics proved to have anti-inflammatory properties that may be beneficial in preventing ileus added to its analgesic actions. The lidocaine patch evaluated in many types of pain with promising results. The study try to evaluate the patch in perioperative field as a more simple and safe technique than the intravenous route.

ELIGIBILITY:
Inclusion Criteria:

* female undergoing elective gynecologic surgery

Exclusion Criteria:

* known allergy to lidocaine,
* respiratory or cardiac dysfunction, arrhythmia, treatment with antiarrhythmic drugs,
* inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* hepatic, renal
* chronic use of analgesics or corticosteroids

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female for laparoscopic gynecology
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain VAS scores at rest and during coughing were recorded postoperatively | 24 hours
  To determine if lidocaine patch is superior to placebo as an adjunctive therapy for acute postoperative pain. Average pain score in women at 24 hours postoperatively. Measured using a Visual Analog Scale (VAS), a scale which measures pain from 0 to 100 with 0="no pain" and 100="the worst pain you have ever felt".

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No